CLINICAL TRIAL: NCT04558372
Title: Genosvid Diagnostic Test for Early Detection of COVID-19: UGM Electronic-Nose Innovation for Indonesia
Brief Title: Genosvid Diagnostic Test for Early Detection of COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, dr. Dian K. Nurputra, M.Sc, Ph.D, SpA, MD(Paed), M.Sc, Ph.D, Gadjah Mada University
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 1.6/2020
Record Dates: First submitted 2020-09-20; First posted 2020-09-22 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: COVID-19
Keywords: COVID-19; diagnosis; electronic nose
MeSH Terms: conditions — COVID-19; Disease

STUDY DESIGN:
Intervention Model Description: 3 groups:
  1. COVID-19 patients
  2. non COVID-19 patients
  3. suspected COVID-19 patients
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The person who operates breath test is blinded to the results of swab. The swab taker is blinded to the result of breath sample. The patients also do not know the results of the interpretation of the breath sample. Patients will receive information on the results of the oro/ nasopharyngeal swab in accordance with the COVID-19 health service standards. The final data processor is also blinded to the results of nose and throat swabs. The breath sampling data is saved in graphic form which interpretation will be carried out later by the data processor at the final stage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1- 43 COVID-19 patients (Experimental): COVID-19 patients breath normally via disposable non-rebreathing mask
  Interventions: Other: exhaled breath sampling
- Group 2- 40 non COVID-19 patients (Experimental): Non COVID-19 patients breath normally via disposable non-rebreathing mask
  Interventions: Other: exhaled breath sampling
- Group 3- suspected COVID-19 patients (Experimental): The participants breath normally using a mask for 2 times then they are asked to inhale and exhale in a forced expiratory volume through an e-nose tube connected to the Hepa-filter at the inlet.
  Interventions: Other: exhaled breath sampling

INTERVENTIONS:
Other: exhaled breath sampling — The participants breath through non-rebreathing mask until the reservoir bag is full. The reservoir bag is connected to Hepa-filter at one side, and another side of Hepa-filter is connected to the electronic-nose (Genosvid) device.
  Other Names: GENOSVID portable exhaled breath sampling
  Arms: Group 1- 43 COVID-19 patients
Other: exhaled breath sampling — The participants breath through non-rebreathing mask until the reservoir bag is full. The reservoir bag is connected to Hepa-filter at one side, and another side of Hepa-filter is connected to the electronic-nose (Genosvid) device.
  Other Names: GENOSVID portable exhaled breath sampling
  Arms: Group 2- 40 non COVID-19 patients
Other: exhaled breath sampling — The participants breath normally using a mask for 2 times then they are asked to inhale and exhale in a forced expiratory volume through an e-nose tube connected to the Hepa-filter at the inlet.
  Other Names: GENOSVID portable exhaled breath sampling
  Arms: Group 3- suspected COVID-19 patients

SUMMARY:
Electronic-nose had been used to diagnose other infectious lung diseases, such as tuberculosis. Universitas Gadjah Mada has developed an electronic-nose device which is easy-to-use, portable, and can be manufactured at a low price. Here the investigators test the electronic-nose to diagnose COVID-19 in Indonesia.

DETAILED DESCRIPTION:
The validation of device is conducted to 43 confirmed COVID-19 patients and 40 confirmed COVID-19 negative patients from Bhayangkara Hospital, RSLKC Bambalipuro in Yogyakarta Special Region, Indonesia.

Afterwards, patients with symptoms suggesting COVID-19 will be recruited using multicentre consecutive sampling. The minimum number of participants required is 1460 subjects. The study use a triple-blind design where the research subjects, breath sample takers, and sample examiners did not know the results of each sampling that had been done. The final data processor was also blinded to the results of nose and throat swabs. The breath sampling data is saved in graphic form which interpretation will be carried out later by the data processor at the final stage.

This study population involve children and adults who come to the COVID-19 outpatient clinic in each participating hospital with a diagnosis of suspected COVID-19 infection. All patients remain in the setting under medical service in accordance with the standard operating procedure (SOP) and clinical practice guidelines (CPG) protocols for handling patients with suspected COVID-19. The patients underwent nasal and oropharyngeal swabs according to the COVID-19 outpatient CPG.

The participants will be asked about symptoms that they have, such as fever, fatigue, dry cough, stuffy/ runny nose, sore throat, myalgia, shortness of breath, and diarrhea. Afterwards, they will be asked to breathe normally using a mask for 2 times, then inhale and exhale in a forced expiratory volume to an air collecting bag that later is connected to the e-nose machine via a HEPA-filter. The performance of breath test will be compared with the performance of symptoms with the reference of RT-PCR results. In addition, participants' demographic and clinical data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with COVID-19, non COVID-19, and suspected COVID-19 infection, based on the results of anamnesis, physical examination, laboratory, X-rays and rapid tests.
* Able to produce samples for RT-PCR examination.
* Agree to participate (sign informed consent). For children, informed consent are obtained from the parents. For adolescent patients, accent consent is asked.
* Patients who do not need oxygen therapy supplementation in the form of mask-type or ventilator. Patients who use oxygen supplementation with nasal cannula are still included as study participants.

Exclusion Criteria:

* Unable to breath deeply due to difficulty breathing due to complications of COVID-19 or other diseases
* The quality of the breath do not meet the standard interpretation of the instrument sensor curve (breath sampel is declared invalid).

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1999 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of electronic nose signal in COVID-19 | 2 years
  sensitivity, specificity, positive predictive value, negative predictive value of electronic nose signal in diagnosing COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Dian K. Nurputra, MD(Paed), M.Sc, Ph.D, Principal Investigator — Faculty of Medicine, Public Health and Nursing Universitas Gadjah Mada; Kuwat Triyana, Prof, Dr.Eng, MSi., Study Chair — Faculty of Mathematics and Natural Sciences Universitas Gadjah Mada
Locations (8):
- Indonesia (8):
  - RS Bhayangkara Tk I R.Said Soekanto, Jakarta
  - Saiful Anwar, Malang
  - Dr Sardjito Hospital, Yogyakarta
  - Bambanglipuro Hospital, Yogyakarta
  - Bhayangkara Tk III Polda DIY, Yogyakarta
  - RS Akademik UGM, Yogyakarta
  - RSPAU Hardjolukito, Yogyakarta
  - RST Tk III Dr Soetarto, Yogyakarta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hidayat SN, Julian T, Dharmawan AB, Puspita M, Chandra L, Rohman A, Julia M, Rianjanu A, Nurputra DK, Triyana K, Wasisto HS. Hybrid learning method based on feature clustering and scoring for enhanced COVID-19 breath analysis by an electronic nose. Artif Intell Med. 2022 Jul;129:102323. doi: 10.1016/j.artmed.2022.102323. Epub 2022 May 17. PMID 35659391